CLINICAL TRIAL: NCT02296021
Title: Helicobacter Pylori Eradication With Berberine Hydrochloride,Esomeprazole,Amoxicillin and Clarithromycin Versus Bismuth,Esomeprazole,Amoxicillin,and Clarithromycin: a Randomized,Open-label, Non-inferiority, Phase Ⅳ Trail
Brief Title: Helicobacter Pylori Eradication With Berberine Quadruple Therapy Versus Bismuth-containing Quadruple Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor/Chief Physician, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20140916-2
Record Dates: First submitted 2014-10-29; First posted 2014-11-20 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Gastritis; Peptic Ulcer; Dyspepsia
Keywords: helicobacter pylori; berberine-containing quadruple therapy; bismuth-containing quadruple therapy
MeSH Terms: conditions — Gastritis; Peptic Ulcer; Dyspepsia | interventions — Berberine; Bismuth; Esomeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- berberine quadruple therapy (Experimental): Berberine 500 mg, esomeprazole 20 mg,amoxicillin 1000 mg, and clarithromycin 500 mg by mouth, twice daily for 14 days.
  Interventions: Drug: Berberine; Drug: esomeprazole; Drug: amoxicillin; Drug: clarithromycin
- bismuth quadruple therapy (Active Comparator): Bismuth 220 mg, esomeprazole 20 mg, amoxicillin 1000 mg, and clarithromycin 500 mg by mouth,twice daily for 14 days.
  Interventions: Drug: Bismuth; Drug: esomeprazole; Drug: amoxicillin; Drug: clarithromycin

INTERVENTIONS:
Drug: Berberine — Berberine-containing quadruple therapy group: given for 14 days at a dose of berberine 100 mg 5 tablets BID, esomeprazole 20 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID.
  Arms: berberine quadruple therapy
Drug: Bismuth — Bismuth-containing quadruple therapy group: given for 14 days at a dose of colloidal bismuth tartrate capsule 55 mg 4 capsules BID, esomeprazole 20 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID.
  Other Names: Bitnal; colloidal bismuth tartrate capsule
  Arms: bismuth quadruple therapy
Drug: esomeprazole — Esmeprazole 20mg 1tablet BID plus amoxicillin 500 mg 2 capsules BID, clarithromycin 500 mg 1 tablet BID, and colloidal bismuth tartrate capsule 55 mg 4 capsules BID or berberine 100 mg 5 tablets BID as a dose given for bismuth-containing quadruple therapy or berberine-containing quadruple therapy.
  Other Names: Nexium
Drug: amoxicillin — Amoxicillin 500 mg 2 capsules BID plus esmeprazole 20mg 1tablet BID, clarithromycin 500 mg 1 tablet BID, and colloidal bismuth tartrate capsule 55 mg 4 capsules BID or berberine 100 mg 5 tablets BID as a dose given for bismuth-containing quadruple therapy or berberine-containing quadruple therapy.
  Other Names: Amoxy ( Uni-Amocin )
Drug: clarithromycin — Clarithromycin 500 mg 1 tablet BID plus amoxicillin 500 mg 2 capsules BID, esmeprazole 20mg 1tablet BID, and colloidal bismuth tartrate capsule55 mg 4 capsules BID or berberine 100 mg 5 tablets BID as a dose given for bismuth-containing quadruple therapy or berberine-containing quadruple therapy.

SUMMARY:
This study aims at evaluating efficacy and safety of berberine-containing quadruple therapy(berberine, esomeprazole, clarithromycin and amoxicillin) versus bismuth-containing quadruple therapy (bismuth,esomeprazole,clarithromycin and amoxicillin) in H. pylori eradication. It is hypothesized that berberine-containing quadruple therapy is non-inferior to bismuth-containing quadruple therapy. Patients with confirmed H. pylori positive status will be randomized to one of the treatments described above. At week 2 and 6 follow-up visits, a urea breath test(UBT) will be performed to confirm eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 28 days and subjects eligibility will be evaluated after informed consent signature. Endoscopy and Urea Breath test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 12 and 14.

Follow-up: includes two visits. approximately 14 days of treatment and 28 days after the end of treatment. Eradication of H. Pylori will be confirmed through urea breath test(UBT).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70,both gender.
2. Patients with upper gastrointestinal symptoms and with documented H.pylori infection.
3. Patients are willing to receive eradication treatment.
4. Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

1. Patients are excluded if they have previously used antibiotics to eradicate adequately recorded infection with H. pylori.
2. Contraindications to study drugs.
3. Substantial organ impairment, severe or unstable cardiopulmonary or endocrine disease.
4. Constant use of anti-ulcer drugs ( including taking proton-pump. inhibitors(PPI) within 2 weeks before the [13C] urea breath test), antibiotics or bismuth complexes (more than 3 times /1 month before screening)
5. Pregnant or lactating women.
6. Underwent upper gastrointestinal Surgery.
7. Patients with Barrett esophageal or highly atypical hyperplasia, have symptom of dysphagia.
8. Evidence of bleeding or iron eficiency anemia.
9. A history of malignancy.
10. Drug or alcohol abuse history in the past 1 year.
11. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
12. Enrolled in other clinical trials in the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative [13C] urea breath test 28 days after the end of eradication.

SECONDARY OUTCOMES:
symptoms effective rates | 14 days of treatment, and 28 days after treatment
  Evaluation effective rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment.
  Symptom effective rate =（total score before treatment - total score after treatment）/total score before treatment x 100%. Total score = frequency + severity.
  Frequency score is calculated by all the frequency of heartburn,reflux,abdominal pain,and flatulence. Severity is accumulated by the degree of symptoms described above,which is divided to 4 degree as 0 presenting none,and 3 presenting most severe.
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache,dizziness,skin rash,other gastrointestinal disorders,pyrexia,cough and back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, Ph. D, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi’an, Shanxi, China